CLINICAL TRIAL: NCT05039723
Title: Combination Treatment With Xeomin, Radiesse, and Belotero for Improvement in Photoaging and Skin Quality
Brief Title: Xeomin, Radiesse, and Belotero Facial/Neck Rejuvenational
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Main Line Center for Laser Surgery (Other)
Collaborators: Merz North America, Inc. (Industry)
Responsible Party: Principal Investigator, Eric Bernstein, MD, Physician, Main Line Center for Laser Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Merz IIT7600
Record Dates: First submitted 2021-09-01; First posted 2021-09-10 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Photoaging
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Treatment with Xeomin, Radiesse, and/or Belotero
  Interventions: Drug: Radiesse, Xeomin, Belotero

INTERVENTIONS:
Drug: Radiesse, Xeomin, Belotero — Rejuvenation with Radiesse, Xeomin, Belotero

SUMMARY:
The purpose of this study is to determine the improvement in signs of photoaging and subject satisfaction after combination, global facial and/or neck treatment with IncobotulinumA (Xeomin), HA (Belotero) and/or calcium hydroxyapatite (Radiesse+, Radiesse Classic). All products will be used on-label FDA-cleared indications.

DETAILED DESCRIPTION:
Facial and neck aging is multifactorial, resulting from changes in anatomical aspects combined with changes in the skin integrity. The 5 key signs of photoaging will be evaluated both objectively and subjectively including: fine lines and wrinkles, enlarged pores, sagging skin, pigmentation and redness/flushing. These aspects of the aging face are often bothersome to patients who seek aesthetic treatments for correction.

Injectables, including IncobutolinumtoxinA, hyaluronic acid (HA), and calcium hydroxyapatite, have grown in popularity over the past decade due to their safety profiles, favorable results, and longevity. IncobutolinumtoxinA allows for correction of rhytides, while HA and calcium hydroxyapatite allow for lifting, contouring, and overall re-volumization. Further, calcium hydroxyapatite effectively restores volume and can improve skin texture through its biostimulatory effects, which have been well studied in the literature. Through inducing collagen formation in the skin, calcium hydroxyapatite can also improve skin quality and thickness. In contrast to volumization effects, the overall improvement in skin quality has not been as well studied. Further, it has been observed by patients and physicians that global treatment with toxins and fillers can produce a better result in skin texture than each agent on its own.

This study will consist of one treatment visit for global facial treatment using toxin and fillers (Xeomin, Radiesse+, Radiesse Classic, Belotero Balance) to enhance signs of facial photoaging and appearance.

This clinical investigation is a prospective study consisting of a screening/treatment visit and 3 follow-up visits. A total of 20 patients will be recruited. Following informed consent and screening, each eligible subject will be photographed with the Canfield Visia system. They will be treated at Baseline Visit (Day 0) with Xeomin, Belotero Balance, Radiesse+, and/or Radiesse Classic. Determination of which facial and/or neck areas to be treated will be made after assessment by the investigator and discussion with the patient. All products will be used on-label in their FDA-cleared manner. Post-treatment, patients will be instructed to apply ice to all areas for 3-5 minutes immediately afterwards.

The patient will return at post-treatment months 1 and 3 for GAIS and FACE-Q Subject Satisfaction and photography with the Canfield Visia system. A blinded independent evaluator will evaluate the baseline and post-treatment photographs on a 5-point scale for fine lines and wrinkles, enlarged pores, redness, flushing, pigmentation, and sagging skin.

ELIGIBILITY:
Inclusion Criteria:

* Age >21
* No toxin treatment in last 3 months
* No filler treatment in last 3 months
* Glogau facing aging scale >=1

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Allergy to prior Radiesse, Belotero, Xeomin products
* History of any facial nerve palsy (ie. Bell's Palsy)

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
FACE-Q Subject Satisfaction | 3 months

SECONDARY OUTCOMES:
Global Assessment Investigator Scale | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kachiu Lee, MD, Study Director — Main Line Center for Laser Surgery; Eric Bernstein, MD, Principal Investigator — Main Line Center for Laser Surgery
Locations (1):
- Main Line Center for Laser Surgery, Ardmore, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No